CLINICAL TRIAL: NCT05256667
Title: Comparison Between Root Canal Treatment in Single and Two Visits, With and Without the Use of Intracanal Dressing, in Periradicular Repair in Teeth With Apical Periodontitis: Double-blinded, Controlled Randomized Trial
Brief Title: Comparison Between RCT in Single and Two Visits, With and Without Intracanal Dressing, in Apical Repair
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2021-12-04; First posted 2022-02-25 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-02

CONDITIONS: Teeth, Endodontically-Treated; Tooth, Nonvital; Periapical Periodontitis, Chronic Nonsuppurative; Periapical Granuloma
Keywords: tooth, nonvital
MeSH Terms: conditions — Tooth, Nonvital; Periapical Granuloma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Root canal treatment in single visit - RCT-SV (Other): Group 1- RCT-SV: Endodontic treatment in a single visit using chemomechanical preparation (rotary NiTi instruments, 5.25% NaOCl, 17% EDTA) and passive ultrasonic irrigation (PUI), followed by obturation (gutta-percha and epoxy resin-based sealer) and final restoration (composite resin).
  Interventions: Combination Product: RCT-SV
- Root canal treatment in two visits with intracanal dressing - RCT-TVWD (Other): Group 2- RCT-TVWD: Endodontic treatment in two visits using chemomechanical preparation (rotary NiTi instruments, 5.25% NaOCl, 17% EDTA) and passive ultrasonic irrigation (PUI), followed by intracanal dressing (calcium hydroxide powder, CPMC, glycerine) and temporary restoration (glass ionomer cement) for 7 days. After 7 days, an identical chemomechanical preparation on visit 2 will be performed, followed by obturation (gutta-percha and epoxy resin-based sealer) and final restoration (composite resin).
  Interventions: Other: RCT-TVWD
- Root canal treatment in two visits without intracanal dressing - RCT-TVWOD (Other): Group 3- RCT-TVWOD: Endodontic treatment in two visits using chemomechanical preparation (rotary NiTi instruments, 5.25% NaOCl, 17% EDTA) and passive ultrasonic irrigation (PUI), followed by temporary restoration (glass ionomer cement) for 2 days, without intracanal dressing. After 2 days, an identical chemomechanical preparation on visit 2 will be performed performed, followed by obturation (gutta-percha and epoxy resin-based sealer) and final restoration (composite resin).
  Interventions: Other: RCT-TVWOD

INTERVENTIONS:
Combination Product: RCT-SV — Group 1- Endodontic treatment in a single visit using chemomechanical preparation and passive ultrasonic irrigation, followed by obturation and final restoration.
  Arms: Root canal treatment in single visit - RCT-SV
Other: RCT-TVWD — Group 2- Endodontic treatment in two visits using chemomechanical preparation and passive ultrasonic irrigation, followed by intracanal dressing and temporary restoration for 7 days. After 7 days, an identical chemomechanical preparation on visit 2 will be performed, followed by obturation and final restoration.
  Arms: Root canal treatment in two visits with intracanal dressing - RCT-TVWD
Other: RCT-TVWOD — Group 3- Endodontic treatment in two visits using chemomechanical preparation and passive ultrasonic irrigation, followed by temporary restoration for 2 days, without intracanal dressing. After 2 days, an identical chemomechanical preparation on visit 2 will be performed, followed by obturation and final restoration.
  Arms: Root canal treatment in two visits without intracanal dressing - RCT-TVWOD

SUMMARY:
This is a randomized, prospective, double-blind, controlled clinical trial designed to evaluate 3 distinct clinical approaches used during endodontic therapy: Group 1- Root canal treatment in single visit (RCT-SV); Group 2- Root canal treatment in two visits with intracanal dressing (RCT-TVWD); Group 3- Root canal treatment in two visits without intracanal dressing (RCT-TVWOD). A total of 210 adult patients ages 18 to 60 years, with at least one tooth diagnosed with asymptomatic apical periodontitis and periradicular lesion will be randomized and will undergo one of the types of clinical approaches during endodontic therapy. Patients' postoperative pain levels will also be recorded in periods of 24, 48, 72 hours and 7 days. Subsequently, clinical findings and long-term follow-up evaluations, with periradicular repair will be performed by periapical radiograph and computed tomography (cone-beam) at 6th, 12th and 24th months.

DETAILED DESCRIPTION:
All patients will voluntarily seek endodontic treatment in the Brazilian Unified Health System in the cities of Itabuna, in the State of Bahia, in Goiânia, in the State of Goiás, Brazil. After an assessment of eligibility and informed consent, patients will be randomly assigned to one of 3 clinical study groups. Patients who agree to participate in this study will sign an informed consent form. Sample Size: The determination of the sample size will be performed sequentially, with a minimum of 210 statistical units (teeth) to be recruited in the first stage, and the second stage of recruitment will be performed if the selection is insufficient to clinically and radiographically identify valid cases. This sampling will also allow the adjustment of the sample size for the intra-subject correlation of statistical units (teeth). In the first stage, 150 adults aged 18 to 60 years, with at least one tooth diagnosed with asymptomatic apical periodontitis and periradicular lesion with a diameter between 1 and 5 mm, will be recruited. Allocation and blinding: Only examiners can open the envelope to check the group allocation and perform the interventions according to the instructions of this study. As a double-blinded trial, the patients and outcome evaluators will be blinded to the group assignment until the completion of the study. Interventions: In order to treat apical periodontitis, in the first visit, the same endodontic instrumentation protocol will be performed for all teeth randomly divided into the 3 study groups. What will vary will be complementary and additional maneuvers such as the use of ultrasonic activation and intracanal medication between visits of endodontic instrumentation. All endodontic therapy procedures will be performed under a dental microscope, except for anesthesia and rubber dam placement steps.

The study will be conducted in the private offices of two of the co-investigators involved in the study (GMA and VHMC), located in the cities of Itabuna (Bahia) and Goiânia (Goiás), Brazil, respectively. All investigators and examiners are specialists in Endodontics with more than 10 years of clinical experience. They will participate in this randomized clinical trial after receiving adequate training to obtain a comprehensive view of the principles and strategy of the 3 clinical approaches that will be used.

Description: First clinical appointment: The first visit will include the following clinical protocol depending on the study group. For the 3 groups (Group 1, Group 2 and Group 3): (1) Anesthesia and caries removal: After local anesthesia with articaine hydrochloride and epinephrine injection (with 1:200,000 adrenaline), all decayed tissue from the tooth is removed; (2) Isolation and access preparation. The tooth is isolated with a rubber dam, disinfected and the pulp chamber will be completely unroofed; (3) Initial irrigation with 5 ml of 5.25% NaOCl; (4) Root canal preparation: The #10 C-Pilot file will be used to perform the glide path along the length of the tooth on the radiograph, irrigated with 2 ml of 5.25% NaOCl, followed by rotary instrumentation with #15/.03, #25/.04 and #30/.05 NiTi files, initially in the cervical and middle thirds, after which the working length with foraminal locator will be performed. Finally, the instrumentation of the apical third will be performed with the same sequence of NiTi rotary files used previously; (5) The canal will be copiously irrigated in three stages using 10ml of 5.25% NaOCl for each of thirds: cervical, middle and apical, totaling 30ml, followed by a final rinse with 10ml of 5.25% NaOCl stirred with the ultrasonic inserts and 10 ml of 17% EDTA stirred also with ultrasonic inserts. The final rinse will be carried out with 10ml of saline solution. Intracanal dressing: Group 1 will not receive intracanal dressing because it will be concluded in single visit. Group 2 will receive intracanal dressing with Ca(OH)2/CPMC/glycerin paste for a period of 7 days. To restrict bacterial regrowth and supply continued disinfection, the root canal will be filled homogeneously to the working length with Ca(OH)2/CPMC/glycerin paste. The tooth will be shielded with glass ionomer cement (GIC) as a temporary restoration. Group 3 will be without intracanal dressing for a period of 2 days, taking into account that the tooth will be shielded with GIC as a temporary restoration. Obturation: Only for Group 1, the root canals will be filled in the first visit. In this group, a #30/.05 gutta-percha cone and epoxy resin-based sealer with the continuous heat wave technique and a final restoration with composite resin will be used. Second clinical appointment: The second visit will include the following clinical protocol depending on the study group. For the 2 remaining groups (Group 2 and Group 3): (1) Anesthesia and restorative material removal. After local anesthesia with articaine hydrochloride and epinephrine injection (with 1:200,000 adrenaline, all temporary restorative material from the tooth is removed. (2) Isolation and Access. The tooth is isolated with a rubber dam and the root canal will be accessed one more time. Group 2: (1) After 7 days, the intracanal dressing will be removed and the root canal will receive a new chemo-mechanical preparation, identical to the one performed in the first visit, and then it will be filled and permanently restored similarly to Group 1. Group 3: (1) After 2 days, the root canal will receive a new chemo-mechanical preparation, identical to the one performed in the first visit, and then it will be filled and permanently restored similarly to Group 1.

ELIGIBILITY:
Inclusion criteria:

* Patients diagnosed with apical periodontitis in lower molar teeth (first or second molars), the periradicular lesion with a diameter between 1 and 5mm analyzed through the real 1:1 tomographic scale
* Asymptomatic patients
* Patients who spontaneously agree and sign the informed consent form
* Patients in good health
* Patients who are not taking antibiotics and anti-inflammatory drugs

Exclusion criteria:

* Patients with systemic diseases (diabetes, transplants, heart disease, liver failure and kidney failure)
* Immunodepressed patients
* Teeth with extensive coronary destruction that makes direct restoration with composite resin unfeasible
* Calcified teeth
* Teeth with incomplete root formation
* Teeth with persistent exudation
* Teeth with anatomical complexities that prevent endodontic treatment in a single visit
* Teeth recommended for endodontic retreatment
* Teeth with advanced periodontal pocket
* Teeth in which foraminal patency is not obtained

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-10-02 (Actual); Primary Completion 2024-03-28 (Estimated); Study Completion 2024-05-28 (Estimated)

PRIMARY OUTCOMES:
Healing of periradicular lesions by radiographic findings according to periapical Index (PAI) | Long-term follow-up evaluation in 24 months.
  The periapical index (PAI) is a structured scoring system for categorization of radiographic features of apical periodontitis. It is based on a visual scale of periapical periodontitis severity and was built upon a classical study of histological-radiological correlations. It is a five-point ordinal scale as listed below: 1. Normal periapical structures; 2. Small changes in bone structure with no demineralization; 3. Changes in bone structure with some diffuse demineralization; 4. Apical periodontitis with well-defined radiolucent area; 5. Severe apical periodontitis, with exacerbating features.

SECONDARY OUTCOMES:
Patient's postoperative pain using questionnaire | Evaluation of postoperative pain after endodontic treatment completion, an average of 7 days.
  Patients will answer a questionnaire for the analysis of postoperative pain, through the analogue pain scale: (a) No pain; (b) Mild pain; (c) Moderate pain; (d) Severe pain; (e) Intense pain.
Patient's preference regarding the number of clinical visits using questionnaire | Immediately before starting endodontic treatment.
  Data on the patient's preference regarding the number of clinical visits to be planned for the conduction of endodontic treatment, patients will answer their preferences according to hypothetical conditions described in a previously delivered questionnaire: (a) Single visit; (b) Multiple visits; (c) No preference.
Patient's post-treatment satisfaction using questionnaire | Immediately after endodontic treatment completion.
  Post-treatment satisfaction questionnaire will be applied to patients undergoing clinical interventions in a single visit and two visits, using the following criteria: (a) Fully satisfied; (b) Satisfied; (c) Neither dissatisfied nor satisfied; (d) Dissatisfied; (e) Totally dissatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Moderne Odontolgia, Itabuna, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share, protocol, methods, results
Supporting Information: Study Protocol, SAP, CSR
Time Frame: after publication - for 6 months
Access Criteria: Free
URL: http://scholar.google.com

REFERENCES:
- [Derived] Almeida GM, Carvalho VHM, Silva EBP, Cancado MAF, Barroso LS, Queiroz EL, An TL, Ribeiro APD, Carvalho-Junior JR, Leite AF. Periradicular repair after single- and two-visit root canal treatments using ultrasonic irrigant activation and calcium hydroxide dressing of teeth with apical periodontitis: study protocol for randomized controlled trials. Trials. 2023 Jan 12;24(1):23. doi: 10.1186/s13063-022-07030-0. PMID 36635764